CLINICAL TRIAL: NCT05163483
Title: Tucidinostat in Combination With PD-1 Inhibitor and Bevacizumab as Late-line Treatment in Patients With Advanced Esophageal Squamous Cell Cancer, Adenocarcinoma of Esophagogastric Junction and Gastric Adenocarcinoma
Brief Title: Tucidinostat Plus PD-1 Inhibitor and Bevacizumab for Advanced Esophagus Cancer, AEG, Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruihua Xu (Other)
Responsible Party: Sponsor-Investigator, Ruihua Xu, Sun Yat-sen University cancer center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q24
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Squamous Cell Cancer, Adenocarcinoma of Esophagogastric Junction, Gastric Adenocarcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Immune Checkpoint Inhibitors; toripalimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat (chidamide), PD-1 inhibitor （Toripalimab), Bevacizumab (Experimental): Tucidinostat (chidamide), 30mg, po., biw, q3w Toripalimab, 240mg, ivgtt., d1, q3w Bevacizumab, 7.5mg/kg, ivgtt., d1, q3w
  approximately 2 years
  Interventions: Drug: Tucidinostat (chidamide), PD-1 inhibitor (Toripalimab), Bevacizumab

INTERVENTIONS:
Drug: Tucidinostat (chidamide), PD-1 inhibitor (Toripalimab), Bevacizumab — Tucidinostat (chidamide), 30mg, po., biw, q3w Toripalimab, 240mg, ivgtt., d1, q3w Bevacizumab, 7.5mg/kg, ivgtt., d1, q3w
  approximately 2 years
  Other Names: Tucidinostat (chidamide) JS001

SUMMARY:
This Phase II study was designed to assess the efficacy and safety of the combination of PD-1 inhibitor, Tucidinostat (chidamide), a histone deacetylase inhibitor, and bevacizumab in advanced Esophageal squamous cell cancer, adenocarcinoma of esophagogastric junction, Gastric adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤ 75 years
2. Histologically or cytologically confirmed Esophageal squamous cell cancer, adenocarcinoma of esophagogastric junction and Gastric adenocarcinoma, unresectable, recurrent or metastatic disease.
3. Can provide at least 5 pieces of pathological section or fresh tumor tissue
4. Eastern Collaborative Oncology Group (ECOG) ≤ 1.
5. ≤2 systemic chemotherapy for advanced disease (total number of treatment lines for advanced disease ≤4).
6. Patients who have previously used PD-1 antibodies, PD-L1 antibodies, PD-L2 antibodies, or CTLA-4 antibodies (or any other antibodies acting on T cell co-stimulation or checkpoint pathways) or require a duration of ≥16 weeks;
7. Adequate organ function.
8. Life expectancy is more than 3 months.
9. For females of child bearing potential, a negative urine or serum pregnancy test result within 3 days before study treatment.
10. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Allergies to any monoclonal antibody or Tucidinostat preparation have been known, and hypersensitivity reactions of more than 3 levels have occurred
2. Previously received immunotherapy and had grade 3 or above immune-related adverse events.
3. Previously received histone deacetylase inhibitors,or toripalimab, or angiogenesis inhibitors.
4. Subjects with any active, known or suspected autoimmune disease or history of autoimmune disease.
5. Known active CNS metastases and/or carcinomatous meningitis.
6. Received a live vaccine within 4 weeks of the first dose of study medication.
7. Major surgery received or severe traumatic injury, fracture, or ulcer occurred within 4 weeks of the first dose of study medication.
8. Pregnant or lactating female.
9. Uncontrolled clinically significant systemic diseases, including active infection, unstable angina, angina occurred within 3 months,≥ NYHA II congestive heart failure, myocardial infarction occurred within 6 months, severe arrhythmia, liver, kidney, or metabolic disease.
10. Participate in other clinical trials currently or within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Time from treatment until disease progression or death
Disease Control Rate （DCR） | 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and stable disease（SD）
Duration of Response（DoR） | 2 years
  Time from the achievement of a response to progression
Overall survival(OS) | 3 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China